CLINICAL TRIAL: NCT03651895
Title: Metformin to Reduce Airway Glucose in COPD Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18SM4819; 2018-001755-12 (EudraCT Number)
Record Dates: First submitted 2018-08-02; First posted 2018-08-29 (Actual); Results first posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group (Active Comparator): Metformin 500mg/1g bd
  Interventions: Drug: Metformin
- Placebo Group (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — The Drug was administered 500 mg twice daily for one week and increased to 1g twice daily for the reminder of the 3 months.
  Arms: Treatment Group
Drug: Placebo — Placebo
  Arms: Placebo Group

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is the 4th leading cause of death worldwide and affects 1.2 million people in the UK, costing the NHS >£800 million annually. COPD patients are more susceptible to bacterial infections and both chronic and acute infections are common. COPD patients with chronic lung bacterial infection have worse quality of life, faster disease progression, more symptoms and frequent exacerbations. Acute infections are the main cause of COPD exacerbations which cause COPD patients to become acutely unwell and often result in hospitalisation especially in the winter. Antibiotics are frequently used to treat COPD exacerbations and this contributes to the development of antibiotic resistance. Therefore there is a need to develop antibiotic-independent approaches to reducing or preventing bacterial infection in COPD.

The investigators have carried out work in in animal studies and in humans showing that there is a link between high levels of glucose in the lung and bacterial lung infection. Levels of glucose in the lung are higher in COPD patients compared with people without COPD. These higher glucose levels support greater bacterial growth probably because glucose is a nutrient for bacteria. Therefore reducing airway glucose has the potential to inhibit bacterial growth in COPD patients.

In animal studies the investigators have demonstrated that the diabetic drug metformin decreases airway glucose and bacterial growth. The investigators wish to determine if metformin can achieve the same effects in COPD patients. Metformin is safe and cheap, and has been extensively used in COPD patients with diabetes with an excellent safety record. The primary aim of this study will be to determine whether metformin reduces lung glucose in a small group of non-diabetic COPD patients. If it demonstrates that metformin reduces lung glucose concentrations it will justify a larger clinical trial of metformin as a treatment for COPD.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is the 4th leading cause of death worldwide and affects 1.2 million people in the UK, costing the NHS >£800 million annually. COPD patients are more susceptible to both chronic and acute bacterial infections. Patients with chronic lung bacterial infection have worse quality of life, faster disease progression, more symptoms and frequent exacerbations. Acute infections are the main cause of acute COPD exacerbations which cause COPD patients to become acutely unwell and often result in hospitalisation especially in the winter. Bacteria are detected in 50-60% of COPD exacerbations. Antibiotics are frequently used to treat COPD exacerbations and this contributes to the development of antibiotic resistance. Therefore any intervention that prevents or reduces bacterial infection in COPD, especially if it is not an antibiotic, will have major benefits for COPD patients, the NHS and for society as a whole.

It is likely that there are many reasons why COPD patients are more susceptible to bacterial infections. From experimental work the investigators have carried out one of the reasons may be high glucose concentrations in the lung.

In healthy lungs glucose levels are kept low and this may be a mechanism that inhibits bacterial growth by depriving them of an essential nutrient. In animal studies the investigators have demonstrated that when levels of glucose in the lung are high, bacterial lung infection is more common. The investigators measured lung glucose concentrations in COPD patients and found that they are higher compared with people without COPD. COPD patients with higher levels of glucose also had more bacteria in their lungs and sputum samples from COPD patients with higher glucose concentrations supported greater bacterial growth in the laboratory.

Therefore this study was the first to link elevated glucose in the lung to bacterial infection in COPD. Therefore reducing airway glucose has the potential to inhibit bacterial growth in COPD patients.

Study Design The proposed study will be a randomised, double-blinded, placebo-controlled, cross-over study of metformin in COPD patients. The primary outcome will be sputum glucose after 3 months' treatment with metformin compared with sputum glucose in those taking placebo. In order to account for potential withdrawals 40 subjects will be recruited.

Study Procedures Potential participants will attend for a screening visit where they will have a full medical history, a physical examination and spirometry carried out to confirm the diagnosis of COPD. A blood test will also be done to measure kidney and liver function and blood glucose to exclude undiagnosed diabetes, kidney disease or liver disease.

If they fulfil the entry criteria and consent to taking part in the study they will have a baseline visit prior to being randomised.

The baseline visit will include:

1. Physical examination and measurement of vital signs
2. Completion of quality of life (St George's Respiratory Questionnaire (SGRQ)) and symptom questionnaires (COPD Assessment Test (CAT))
3. Collection of samples. The samples collected will include blood samples, nose samples collected using nasal synthetic absorption matrix (SAM) strips and induced sputum.

After baseline assessment, subjects will either be commenced on metformin (500mg twice a day after meals) or placebo for 3 months during which time the participants will have monthly visits. At these visits the same assessments and sampling as the baseline will be carried out, together with collection of data regarding exacerbations and adverse events. Following a 2 week washout period the subjects will crossover to the other study arm for another 3 months and follow the same study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 75 years
* Clinical diagnosis of COPD confirmed with spirometry (Post-bronchodilator FEV1/FVC <70%).
* Smoking history >15 pack years
* Absence of infection >8 weeks prior to study entry
* No use of antibiotics and/or oral corticosteroids >8 weeks prior to study entry
* Able to understand and consent to the study procedures

Exclusion criteria:

* Diabetes including diabetes diagnosed at screening
* History of hepatic or renal impairment or diagnosed on screening bloods
* Patients already taking metformin irrespective of indication
* Known allergy or hypersensitivity to metformin
* Pregnancy or breastfeeding
* Any other significant medical condition likely to interfere with the study
* Unable to provide informed consent
* Excessive alcohol intake (>21 units/week)
* BMI < 18.5kg/m2

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Johnston, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Respiratory Research Unit, St Mary's Hospital, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall treatment time 6 months (2 milestones at 1 and 3 months)
Pre-assignment Details: 14 participants were enrolled but 11 withdrew for lower/upper respiratory tract infections (LRTI/URTI) Cough and Vomiting. At 3 months there was a washout and a crossover thereafter.
Groups:
- Metformin First (Before Crossover), Placebo Second (After Crossover); Placebo First (Before Crossover), Metformin Second (After Crossover): Metformin 500 milligrams (mg)/1 gram (g) twice daily.
  Metformin: 500mg twice daily was administered for one week and increased to 1g twice daily for the reminder of the 3 months.
  Placebo
  Placebo: The drug was administered with the same regime as the metformin.
Period: First Drug Assignment
Arm/Group | Metformin First (Before Crossover), Placebo Second (After Crossover) | Placebo First (Before Crossover), Metformin Second (After Crossover)
Started | 7 | 7
1 Month | 6 | 6
3 Months | 3 | 2
Completed | 3 | 2
Not Completed | 4 | 5
Not completed — Adverse Event | 4 | 5
Period: Second Drug Assignment - Crossover
Arm/Group | Metformin First (Before Crossover), Placebo Second (After Crossover) | Placebo First (Before Crossover), Metformin Second (After Crossover)
Started | 2 | 3
1 Month | 2 | 2
Completed | 1 | 2
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Treatment Group & Placebo Group: Placebo
  Or
  Metformin 500mg/1g bd
  Metformin: The Drug was administered 500 mg twice daily for one week and increased to 1g twice daily for the reminder of the 3 months.
Arm/Group | Treatment Group & Placebo Group
Number analyzed (Participants) | 14
Age, Customized [Mean (Full Range); unit: years]
  Age | 67.9 [53 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 12
  Others | 2
Region of Enrollment [Number; unit: participants]
  United Kingdom | 14
Forced Expiratory Volume in One Second (FEV1) Percentage (%) Predicted [Mean (Standard Deviation); unit: Percentage(%) predicted] | 68.2 (17.8)
Forced Vital Capacity (FVC) Percentage (%) Predicted [Mean (Standard Deviation); unit: Percentage (%) predicted] | 100.3 (15.1)
Peak Expiratory Flow (PEF) Percentage (%) Predicted [Mean (Standard Deviation); unit: Percentage (%) predicted] | 65.4 (22.8)
COPD Assessment Test (CAT) [Mean (Standard Deviation); unit: Score on a scale] | 15.4 (9.3)
St George's Respiratory Questionnaire (SGRQ) [Mean (Standard Deviation); unit: Score on a scale] | 41.8 (16.2)
Sputum Glucose Concentration [Median (Inter-Quartile Range); unit: µmol] | 5.3 [0.02 to 18]

OUTCOME MEASURES:

1. Primary Outcome: Sputum Glucose Concentration
Description: The median concentration of glucose in sputum following 3 months treatment with metformin or placebo.
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: µM
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 4 | 4
µM | 68.92 [16.3 to 131.1] | 12.2 [10 to 13]

2. Secondary Outcome: Nasal Glucose Concentrations
Description: The median concentration of glucose in nasal samples following 3 months treatment with metformin or placebo.
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: µM
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 4 | 4
µM | 12.56 [5.92 to 28.28] | 13.5 [6.19 to 27.83]

3. Secondary Outcome: Sputum Bacterial Load
Description: The bacterial load in sputum using qPCR was not measured. Therefore, data were not collected
Time Frame: 3 months
Population: Data were not collected. Participants with infection were excluded from the study.
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Sputum Inflammatory Markers
Description: The median concentration of inflammatory cells and cytokines in sputum was not measured. Therefore, data were not collected.
Time Frame: 3 months
Population: Data were not collected. Participants with infection were excluded from the study.
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Quality of Life Score (COPD Assessment Test)
Description: The COPD Assessment Test (CAT): the CAT features 8 questions ranked from 0-5 with a minimum score of 0 and maximum possible score of 40. Higher scores indicate a greater impact on patient health due to their COPD, a difference of ≥2 is considered meaningful.
  The questionnaire's were completed by every participant at every visit up to 8 times: V1 is at the baseline, then V2-4 are at monthly intervals. V5 is at the baseline after crossing arms -1 month washout, V6-8 are monthly after that.
Time Frame: 1 month
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 8 | 8
Score on a scale | 16.6 [6.4 to 26.8] | 13.2 [3.3 to 23.1]

6. Secondary Outcome: Quality of Life Score (St George's Respiratory Questionnaire)
Description: St George's Respiratory Questionnaire (SGRQ): the SGRQ contains 50 items with a minimum score of 0 and a maximum score of 100. Higher scores indicate a greater impact on quality of life due to COPD and a difference of ≥4 is meaningful
  The questionnaire's were completed by every participant at every visit up to 8 times: V1 is at the baseline, then V2-4 are at monthly intervals. V5 is at the baseline after crossing arms -1 month washout, V6-8 are monthly after that.
Time Frame: 1 month
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 8 | 8
Score on a scale | 42.7 [24.4 to 61] | 36.4 [18.6 to 54.2]

7. Secondary Outcome: Lung Function
Description: FEV1(Forced Expiratory Volume Test) was performed up to 8 times: V1 is at the baseline, then V2-4 are at monthly intervals. V5 is at the baseline after crossing arms -1 month washout, V6-8 are monthly after that.
Time Frame: 1 month
Measure: Median (Inter-Quartile Range); unit: Litres (L)
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 8 | 8
Litres (L) | 69.2 [51 to 87.4] | 66.1 [46.7 to 85.5]

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse events were reviewed at every study visit.
Groups:
- Placebo Group: Placebo
  Placebo: The Drug was administered 500 mg twice daily for one week and increased to 1g twice daily for the reminder of the 3 months.
Arm/Group | Treatment Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 1/14
Other Adverse Events (participants affected / at risk) | 7/14 | 7/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group (N=14) | Placebo Group (N=14)
Exacerbation of COPD with hospitalisation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group (N=14) | Placebo Group (N=14)
Nausea (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Abdominal cramps (Gastrointestinal disorders) | 1 | 0
Lower respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Procedural related adverse event (Respiratory, thoracic and mediastinal disorders) | 1 | 3 — Breathlessness or lightheadedness during sputum induction

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-03): https://cdn.clinicaltrials.gov/large-docs/95/NCT03651895/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-03): https://cdn.clinicaltrials.gov/large-docs/95/NCT03651895/ICF_001.pdf